CLINICAL TRIAL: NCT02222038
Title: Investigation of the Genetic Architecture of Linear Localized Scleroderma (LLS) (Linear Morphea) by Whole Exome Sequencing. A Tailored Approach to Test the Hypothesis That LLS is a Genetic Mosaic Condition
Brief Title: Genetic Variants in Linear Localized Scleroderma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KISPI-UZH-LLS-2014
Record Dates: First submitted 2014-07-21; First posted 2014-08-21 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Morphea
MeSH Terms: conditions — Scleroderma, Localized

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- skin biopsy (Other): 4mm punch biopsy
  Interventions: Other: skin biopsy

INTERVENTIONS:
Other: skin biopsy

SUMMARY:
The purpose of this study is to investigate the genetic architecture of Linear Localized Scleroderma (LLS) (linear morphea) by whole exome sequencing.

DETAILED DESCRIPTION:
At present the etiology of LLS is unknown, but a genetic background is suspected. Although LLS clearly classifies as a mosaic disorder, its genetics and protein machinery remain to be understood.

We are going to use a tailored approach to identify the genetic factors of LLS. In the first phase of the study we will investigate the genetic architecture in LLS. WES will analyze whole protein coding DNA in skin samples of 50 consenting LLS patient. The aim is to identify the key genes associated with LLS. In the second phase of the study subsequent functional experiments will be performed. Based on the identified candidate genes, knockdown and overexpression models will be created with relevant cell lines (fibroblasts) to identify the biological consequences and confirm the functional relevance of the identified genetic mutations in LLS. Further the protein network active in LLS will be investigated (proteomic analysis).

The described basic genetic studies combined with functional experiments will lay the groundwork for treatment trials to provide possibly novel treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥ 5 years of age with well phenotyped LLS
* Affecting their head and / or face "termed " en coup de sabre " type LLS or Hemiatrophia faciei or Parry-Romberg syndrome, with or without therapy
* Affecting any site of the body except the head or face, with or without therapy

Exclusion Criteria:

* Patients with signs of systemic scleroderma
* Patients with localized scleroderma (morphea) other than the linear type ("plaque-type", "morphea profunda", "generalized morphea") Patients with diagnosed gadolinium induced scleroderma Patients with post-irradiation scleroderma Patients with missing consent

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-08; Primary Completion 2017-10 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
number of key genes /number of mutations in LLS (localized linear scleroderma) | 24-30 months

SECONDARY OUTCOMES:
the investigation of the protein network of the identified key genes in order to assess their biological function and their relevance in the pathogenesis of LLS. | 24-30 months

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Weibel, MD, Principal Investigator — Department Pediatric Dermatology University Children's Hospital Zurich
Locations (2):
- Switzerland (2):
  - University Children's Hospital, Department of Pediatric Dermatology, Zurich
  - University Hospital, Department of Dermatology, Zurich